CLINICAL TRIAL: NCT01234272
Title: Comparison of the Analgesic Effect Between Intrathecal Morphine and IV-fentanyl Patient Controlled Analgesia (ITM-IVPCA) and Epidural PCA (PCEA) in Patients Undergoing Gastrectomy -Randomized Allocation Study-
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Bon-Nyeo Koo / Associate Professor, Severance Hospital, Department of Anesthesiology & Pain Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2010-0368
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Gastric Cancer
Keywords: patients with; undergoing; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Morphine; Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ITM-IVPCA (Experimental): ITM-IVPCA:intrathecal morphine and IV-fentanyl patient controlled analgesia
  Interventions: Drug: morphine
- PCEA (Active Comparator): PCEA:epidural PCA(patient controlled analgesia)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: morphine — ITM-IVPCA: intrathecal administration of 0.3 mg morphine before induction of general anesthesia and application of IVPCA (basal infusion: fentanyl 0.4mcg/kg/hr, bolus: 0.16mcg/kg of fentanyl with a lock out time of 15 min)
  Arms: ITM-IVPCA
Drug: Ropivacaine — PCEA: epidural administration of 5ml 0.2% ropivacaine before induction of general anesthesia and application of PCEA (basal infusion: 5ml 0.2% ropivacaine with fentanyl 0.4 mcg/kg/hr, bolus: 2ml 0.2% ropivacaine with fentanyl 0.16mcg/kg with a lockout time 15min)
  Arms: PCEA

SUMMARY:
The present study was designed to assess analgesic capacity of intrathecal administration of morphine combined with intravenous fentanyl patient-controlled analgesia (ITM-PCA) compared to patient controlled epidural analgesia using fentanyl and repivacaine (PCEA) in patients undergoing gastrectomy. The investigators hypothesized that ITM-PCA would show comparable analgesic effect to PCEA in gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* I or II of preoperative physical status classification by the American Society of Anesthesiologists.
* more than 20 years old.
* undergoing gastrectomy due to gastric cancer.

Exclusion Criteria:

* contraindication to regional anesthesia technique (bleeding diasthesis, sepsis etc) or spine anomaly.
* prior history of abdominal surgery or spine surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Nyeo Koo, MD, Ph.D, Principal Investigator — Severance Hospital, Department of Anesthesia and Pain Medicine
Locations (1):
- Severance Hospital, Seoul, South Korea